CLINICAL TRIAL: NCT00862004
Title: Feasibility of Video-Assisted Thoracoscopic Surgery for Clinical Stage IIIA Non-Small Cell Lung Cancer
Brief Title: Video-assisted Thoracoscopic Surgery for Stage IIIA Non-Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Guangzhou Medical College, the First Affiliated Hospital of Guangzhou Medical College
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FAHG20081202
Record Dates: First submitted 2009-03-13; First posted 2009-03-16 (Estimated); Last update posted 2010-02-02 (Estimated); Status verified 2009-03

CONDITIONS: Non-small Cell Lung Cancer
Keywords: video-assisted thoracoscopic surgery (VATS); systematic node dissection (SND); stage IIIA non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Thoracic Surgery, Video-Assisted

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: VATS — video-assisted thoracoscopic surgery (VATS) major pulmonary resection with systematic node dissection (SND) for clinical stage IIIA non-small cell lung cancer

SUMMARY:
The purpose of this study is to examine the feasibility of video-assisted thoracoscopic surgery (VATS) major pulmonary resection with systematic node dissection (SND) for clinical stage IIIA non-small cell lung cancer. Success is defined as VATS major pulmonary resection with SND without conversion. If success rate over 90%, VATS major pulmonary resection with SND is considered as feasible procedures for clinical stage IIIA non-small cell lung cancer.

DETAILED DESCRIPTION:
Video-assisted or minimally invasive surgery has become the standard approach for many abdominal surgical operations such as cholecystectomy and fundoplication. With respect to the thorax, video-assisted thoracoscopic surgery (VATS) is the accepted technique for biopsy of the lung and pleura and surgical treatment of pneumothorax. A VATS lobectomy with systematic node dissection (SND) for non-small cell lung cancer (NSCLC) has been gradually introduced by many thoracic surgeons since it was first performed in 1995 by McKenna and associates. They reported that the survival rate for stage I lung cancer is similar between lobectomies done by VATS and by thoracotomy. Although minimally invasive surgery certainly sounds good, it is problematic if it decreases patient's safety or the oncological treatment's effect. Hence, the feasibility and safety of SND by VATS remain controversial. In many institutions, the indication for VATS major pulmonary resection is limited to clinical stage I or II. For the application of the procedure to clinical stage IIIA, it remains controversial. Recently, Watanabe et al. did a retrospective study aimed at determining the outcome of patients with cN0-pN2 NSCLC who underwent VATS major pulmonary resection with SND versus the outcome after major pulmonary resection with SND by open thoracotomy. It demonstrated that VATS major pulmonary resection with SND was a feasible approach to management of cN0-pN2 NSCLC without loss of curability. It was unnecessary to convert the VATS approach to thoracotomy in order to do SND even if pN2 disease is revealed during VATS major pulmonary resection. The purpose of this study is to know whether VATS major pulmonary resection with SND for clinical stage IIIA non-small cell lung cancer is possible.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed non-small cell lung cancer (Squamous, adenosquamous, large cell, or poorly differentiated)
* Stage IIIA (T1-3, N2, M0): N2 disease confirmed by any of the following: Mediastinoscopy; Bronchoscopy with fine-needle aspiration or esophagoscopy; or PET scan
* ECOG performance status 0-1
* Hematopoietic: WBC at least 4,000/mm^3; Platelet count at least 100,000/mm^3
* Hepatic: Bilirubin normal; AST/ALT no greater than 1.5 times upper limit of normal (ULN); Alkaline phosphatase no greater than 2.5 times ULN
* Renal: Creatinine clearance greater than 60 ml/min
* Cardiovascular: Cardiac function normal

Exclusion Criteria:

* Severe complications or infections
* Pregnant or breast-feeding women
* Clinically significant heart disease
* Uncontrolled hepatitis, chronic liver disease, or diabetes mellitus
* Another active cancer except properly treated carcinoma in situ of the cervix or basal/squamous cell skin carcinoma

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-12; Primary Completion 2009-08 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
If success rate over 90%, VATS major pulmonary resection with SND is considered as feasible procedures for clinical stage IIIA non-small cell lung cancer (Success is defined as VATS major pulmonary resection with SND without conversion). | 2 month

SECONDARY OUTCOMES:
To evaluate the intraoperative(surgical duration, estimated blood loss) and postoperative variables(mortality, morbidity, chest tube drainage duration, wound pain, hospital stay) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jianxing He, MD, FACS, Study Chair — Department of Cardiothoracic Surgery, the First Affiliated Hospital of Guangzhou Medical College
Locations (1):
- Department of Cardiothoracic Surgery, the First Affiliated Hospital of Guangzhou Medical College, Guangzhou, Guangdong, China

REFERENCES:
- [Result] Watanabe A, Mishina T, Ohori S, Koyanagi T, Nakashima S, Mawatari T, Kurimoto Y, Higami T. Is video-assisted thoracoscopic surgery a feasible approach for clinical N0 and postoperatively pathological N2 non-small cell lung cancer? Eur J Cardiothorac Surg. 2008 May;33(5):812-8. doi: 10.1016/j.ejcts.2008.01.064. Epub 2008 Mar 14. PMID 18342533
- [Result] He J, Yang Y, Chen M. [Lobectomy by video-assisted thoracoscopic surgery]. Zhonghua Wai Ke Za Zhi. 1996 Feb;34(2):76-8. Chinese. PMID 9388326
- [Result] Shao WL, Liu LX, He JX, Yang YY, Chen HZ, Wu ZF, Wei B, Yin WQ, Yang DK. [Bronchial sleeve resection and reconstruction of pulmonary artery by video-assisted thoracic small incision surgery for central lung cancer: a report of 139 cases]. Zhonghua Wai Ke Za Zhi. 2007 Nov 15;45(22):1530-2. Chinese. PMID 18282386